CLINICAL TRIAL: NCT02889718
Title: Anesthesia Feasibility Study With the CONCERT-CL® Station: Administration of Hypnotic in Closed Loop and Administration of Morphine in TCI Mode, at Constant Concentration, After Initial Calibration With a Pupillometer
Brief Title: Anesthesia Feasibility Study With the CONCERT-CL® Station
Acronym: CONCERT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICO-N-2014-07
Record Dates: First submitted 2016-08-25; First posted 2016-09-07 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Cancer; Surgery
MeSH Terms: conditions — Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- anaesthesia with CONCERT-CL® station (Experimental): During the surgery, 3 drugs usually used for anaesthesia will be administered by the CONCERT-CL® station
  Interventions: Device: CONCERT-CL® station; Other: Surgery

INTERVENTIONS:
Device: CONCERT-CL® station — During cancer surgery (surgery > 1 hour), CONCERT-CL® station will be used in accordance with its CE marking to administer anesthetic agents:
  * Port B = open loop: Analgesic
  * Port A = closed loop: Hypnotic
  * Port C = closed loop: Curare
Other: Surgery — Regardless of the type of surgery the patient receives for his cancer, this surgery must be greater than 1 hour.

SUMMARY:
This is a feasibility study of anesthesia in closed loop with the CONCERT-CL® station, on the effect of the hypnotic agent, measured by the bispectral index of the electroencephalogram, to maintain the hypnosis level within the recommended limits for general anesthesia. The analgesic agent is administered in "Target-Controlled Infusion = TCI" and analgesia evaluated by pupillometry.

This is a prospective, open, non-controlled, non-randomized, monocentric study. The main objective is to study the potential contribution of the system in the conduct of anaesthesia, as decision support, for the administration of the hypnotic agent.

Secondary objectives will include hemodynamic stability, and the average concentrations of opioid and hypnotic anesthetic agents evaluated from the pharmacokinetic model.

The study will involve surgical patients scheduled for surgery under general anesthesia for more than 1 (one) hour.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged 18 years old and over
* Surgery of any type programmed for longer than 1 hour
* Anesthesia combining three agents: hypnotic, morphine, curare

Exclusion Criteria:

* minor patient
* pregnant and lactating women
* Known or suspected hypersensitivity to propofol,
* known or suspected hypersensitivity to remifentanil and other fentanyl derivatives,
* known or suspected hypersensitivity to rocuronium and atracurium, preventing the use of the two products.
* peanut allergy, soy, Egg
* neurological disease history with known modification of the electroencephalogram
* severe eye disease, ocular implant, standing diabetes with diabetic retinopathy
* gravis
* pacemakers patient
* surgery whose position is not suitable for a monitoring on the ulnar nave
* general anesthesia associated with regional anesthesia
* Simultaneous use of shortwave therapy or microwave
* Simultaneous use of high frequency surgical apparatus
* 15 patients under supervision or unable to consent
* patient undergoing psychiatric care
* patient in a health or social institution
* emergency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-02-16 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
During anaesthesia, feasibility of administering hypnotic closed loop with CL® CONCERT station | From start of anesthesia until the release of the patient from recovery room
  The evaluation will measure the level of hypnosis during surgery.
  => The performance of the closed loop of the CONCERT-CL® station will be evaluated by studying its overall score (GS).

CONTACTS AND LOCATIONS:
Overall Officials: MAVOUNGOU Philippe, MD, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (1):
- ICO, Saint-Herblain, France

IPD SHARING:
Plan to Share IPD: No